CLINICAL TRIAL: NCT03058497
Title: A Multi-centre Randomised, Double Blind, Placebo-controlled, Parallel Group Trial of the Effectiveness of the Nocturnal Use of a Temperature Controlled Laminar Airflow (TLA) Device (Airsonett®) in Adults With Poorly-controlled, Severe Allergic Asthma
Brief Title: Laminar Airflow in Severe Asthma for Exacerbation Reduction
Acronym: LASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/33/28
Record Dates: First submitted 2017-01-06; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temperature-Controlled Laminar Airflow Device Active (Active Comparator): Temperature-Controlled Laminar Airflow Device
  Interventions: Device: Temperature-Controlled Laminar Airflow Device (Airsonett®)
- Temperature-Controlled Laminar Airflow Device Placebo (Placebo Comparator): Temperature-Controlled Laminar Airflow Device
  Interventions: Device: Temperature-Controlled Laminar Airflow Device (Airsonett®)

INTERVENTIONS:
Device: Temperature-Controlled Laminar Airflow Device (Airsonett®)

SUMMARY:
To ascertain whether home-based nocturnal TLA usage over a 12 month period can reduce exacerbations and improve asthma control and quality of life as compared to placebo, whilst being cost-effective and acceptable to adults with poorly-controlled, severe allergic asthma.

DETAILED DESCRIPTION:
We will include 222 adults, half of whom will be given a TLA device that is working, and the other half will be given a device which has been inactivated (the filtering process will be switched off, although the participants will not be able to tell that this has occurred). Which participant receives the working or deactivated device will be decided by a random process and will be unknown to the researcher and the participant. An engineering team from the manufacturer will install the device in the participants' home at the beginning of the study and be available throughout the study period to deal with any queries.

All participants will continue receiving their usual treatments. Participants will be in the study for 12 months, and will report their asthma attacks to the trial team whenever they occur during this period. In addition, they will visit the trial team 4 times (after 3, 6, 9 and 12 months) to assess their asthma control and quality of life. At the end of the trial, we will invite participants at each site to join a group discussion where researchers will explore the participant's thoughts about the TLA device. At the end of their participation in the trial, all participants who have used the device for more than 6 months, regardless of their initial study group, will be offered the opportunity to keep an active device in their home free of charge for a further four years.

ELIGIBILITY:
Inclusion Criteria:

- A clinical diagnosis of asthma for ≥6 months with either: Airflow variability Airway reversibility Airway hyper-responsiveness

* Requirement for high-dose inhaled corticosteroids (ICS) (≥1000μg/day beclomethasone (BDP) or equivalent
* Poorly controlled asthma demonstrated by BOTH

  ≥2 severe asthma exacerbations, ACQ (7-point) score >1 at Screening Visit 1 and Randomisation Visit 2
* Atopic status
* Exacerbation free
* Able to use the TLA device during sleep on at least five nights per week
* Able to understand and give written informed consent prior

Exclusion Criteria:

* Current smokers or ex-smokers abstinent for <6months
* Ex-smokers with ≥15 pack year smoking history
* Partner who is a current smoker and smokes within the bedroom where the TLA device is installed
* TLA device cannot be safely installed within the bedroom
* Intending to move out of study area within the follow-up period
* Documented poor treatment adherence
* Occupational asthma with continued exposure to known sensitising agents in the workplace
* Previous bronchial thermoplasty within 12 months of randomisation
* Treatment with Omalizumab (anti-IgE) within 120 days of randomisation
* Using long-term oxygen, Continuous Positive Airway Pressure (CPAP) or Non-Invasive Ventilation (NIV)
* Presence of clinically significant lung disease other than asthma, including smoking-related chronic obstructive pulmonary disease (COPD), bronchiectasis associated with recurrent bacterial infection, allergic bronchopulmonary aspergillosis (mycosis), pulmonary fibrosis, sleep apnoea, pulmonary hypertension, or lung cancer,
* Patients currently taking part in other interventional respiratory clinical trials

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Exacerbation frequency | 12 months
  The frequency of severe asthma exacerbations occurring within the 12 month follow-up

SECONDARY OUTCOMES:
Asthma Control | 12 months
  • To assess the impact of nocturnal TLA treatment on asthma control which includes: Current clinical asthma control
Treatment effect on quality of Life | 12 months
  • To ascertain the effect of TLA treatment on quality of life in poorly-controlled severe allergic asthmatic participants and their carers.
  This will be measured via patient questionnaires
Evaluate the device | 12 months
  • To qualitatively evaluate the perceptions, values and opinions of the device to identify potential modifications to improve patient acceptance and to inform future implementation of the device within the NHS setting
  This will be measured by the participants usage via a completed diary over the 12m period.
NHS Costs | 12 months
  To evaluate the impact of TLA treatment on healthcare utilisation and related costs, and its impact on education/work days lost
NHS Costs | 12 months
  To fully assess the cost-effectiveness, both at one-year and over the lifetime of the patient, of nocturnal TLA treatment using a cost-utility analysis to determine the incremental cost per QALY gained

CONTACTS AND LOCATIONS:
Overall Officials: Anoop[ Chauhan, Study Chair — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospital NHS Trust, Portsmouth, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial Website — http://www.asthma-treatment.org.uk/